CLINICAL TRIAL: NCT05480657
Title: AT-1501-I206: An Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of Transplanted Islet Cells and AT-1501 Immunomodulation in Adults With Brittle Type 1 Diabetes
Brief Title: Safety, Tolerability, and Efficacy of Immunomodulation With AT-1501 in Combination With Transplanted Islet Cells in Adults With Brittle T1D
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study withdrawn
Sponsor: Eledon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-1501-I206
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Brittle Type 1 Diabetes Mellitus
Keywords: AT-1501; Type 1 Diabetes; T1D; Islet Cell Transplant; humanized blocking antibody to CD40L; CD40L inhibitor; monoclonal antibody; Glucose Metabolism Diseases; Diabetes Mellitus; Type 1; Endocrine System Diseases; Graft; Metabolic Diseases; Immune System Diseases; Autoimmune Diseases; Hypoglycemia; Hyperglycemia; Brittle T1D; Brittle Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Endocrine System Diseases; Metabolic Diseases; Immune System Diseases; Autoimmune Diseases; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm AT-1501 (Experimental): Single-arm, open-label trial
  Interventions: Biological: AT-1501 IV Infusion; Biological: Isolated cadaveric islet cells

INTERVENTIONS:
Biological: AT-1501 IV Infusion — Investigational study drug
Biological: Isolated cadaveric islet cells — Infusion of human cadaveric islet cells into the portal vein

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of AT-1501 in an immunomodulation regimen in adult patients with T1D undergoing an islet cell transplant.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability and efficacy of transplantation of experimental islet cells as a potential treatment for brittle type 1 diabetes mellitus. It will also assess the safety, tolerability and efficacy of AT-1501 in an immunomodulation regimen in adult patients with brittle T1D undergoing an islet cell transplant. This is a single arm open-label study and up to 6 participants will be recruited at a single center in the United States.

The objectives include:

* To assess the safety and tolerability of transplanted islet cells and immunomodulation with AT-1501, in combination (AT+) with rabbit anti-thymoglobulin (ATG), etanercept and mycophenolate mofetil (MMF/EC-MPS) in adults with T1D undergoing islet cell transplant.
* To assess the efficacy of transplanted islet cells and immunomodulation with AT-1501 in adults with brittle T1D undergoing islet cell transplant.

The duration of treatment may vary from participant to participant and could be up to 2 years. Participants may receive up to 2 islet cell transplants.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years of age
* A diagnosis of T1D ≥5 years with onset of disease at <40 years of age
* Involvement in appropriate diabetes management in accordance with the standard of care, as directed by an endocrinologist or diabetologist with at least 3 clinical evaluations within the 12 months prior to Screening; using an insulin pump or multiple daily injection (MDI) insulin therapy; and, unable to achieve acceptable metabolic control because of the occurrence of unexplained SHEs
* At least 3 unexplained SHEs not secondary to a missed meal or dosing error, in the 12 months prior to Screening
* Glycosylated hemoglobin (HbA1c) level greater than 7% (53 mmol/mol) and less than 9.5% (80 mmol/mol) inclusive
* Absence of stimulated C peptide (< 0.3 ng/mL) in response to a mixed meal tolerance test (MMTT) measured at 60 and 90 minutes after the start of consumption
* Impaired awareness of hypoglycemia (IAH) as defined by a Clarke Score [Clarke 1995] of 4 or more at the time of Screening, during the Screening period, and within the last 6 months prior to the transplant

Exclusion Criteria:

* Any previous solid organ or islet allotransplant
* Body mass index (BMI) >30 kg/m2
* Insulin requirement >1.0 unit/kg/day or <15 units/day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse Events (AE) and Adverse Events of Special Interest (AEoSI) | Accessed from date of transplant through Day 364 post final transplant for approximately 2 years
  Incidence of adverse events
Efficacy - Insulin independence | Date of transplant through Day 364 post- final transplant
  The proportion of participants that become insulin independent at Days 75 and 365 post-first, and final transplant

SECONDARY OUTCOMES:
Efficacy - HbA1c | Date of transplant through Day 364 post-final transplant
  Proportion of participants with HbA1c <7.0% (53 mmol/mol) and free of serious hypoglycemic events (SHEs) from Day 28 to Day 364 post first and final transplant.
Efficacy - Graft failure | Proportion of participants with graft failure at Day 364 post final transplant
  Date of transplant through Day 364 post final transplant
Efficacy - Durability of insulin independence | Date of transplant through Day 364 post final transplant
  The proportion of participants that become insulin independent at Day 364 post-transplant
Efficacy - Durability of insulin independence - long term | 2 and 3 years after discontinuation of AT- 1501
  The proportion of participants that become insulin independent at year 2 and year 3

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Bornstein, MD, Study Director — Eledon Pharmaceuticals
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No